CLINICAL TRIAL: NCT04144829
Title: Platelet-rich Fibrin Versus HIFU in Management of Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intima Clinic (Industry)
Responsible Party: Principal Investigator, Tomasz Basta, Principal Investigator, Intima Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Intima1/2019
Record Dates: First submitted 2019-10-27; First posted 2019-10-30 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Fibrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIFU (Active Comparator): 3 cycles of HIFU treatment in 6-week intervals
  Interventions: Procedure: HIFU
- Fibrin (Active Comparator): 3 cycles of platelet-rich fibrin injection treatment in 6-week intervals
  Interventions: Procedure: Fibrin

INTERVENTIONS:
Procedure: HIFU — Intravaginal HIFU procedure, lengths 1.5, 3 and 4.5 mm - 200, 200 and 100 impulses respectively
  Arms: HIFU
Procedure: Fibrin — Injection of 2ml platelet-rich fibrin from centrifuged for 5 min patient's blood under the urethra
  Arms: Fibrin

SUMMARY:
Aim of the study is to compare effect of High Intensity Focused Ultrasound (HIFU) and platelet-rich fibrin in management of stress urinary incontinence.

It is a randomized prospective study. After assigning to one of the two groups, patients will undergo relevant treatment.

First group will undergo 3 cycles of intravaginal HIFU treatment in 6-weeks interval.

Second group will undergo 3 injections of platelet-rich fibrin under urethra. Before the treatment and after 2, 6 and 12 months after treatment is finished patients will be asked to fill questionaries concerning quality of life ICIQ-UI SF, ICIQ-LUTS, PISQ12, FSFI.

Before each treatment cycle patients will be examined and asked to fill daily micturition plan.

ELIGIBILITY:
Inclusion Criteria:

* stress urinary incontinence of low grade
* separate episodes of urinary incontinence (associated with increase of abdominal pressure)
* no cystocoele or cystocoele POPQ1
* positive cough test when filled bladder

Exclusion Criteria:

* POPQ 2 and more
* patients after urogenital operations or radiation
* neuromuscular, hematologic, autoimmune, uncontrolled psychiatric diseases
* uncontrolled diabetes
* pregnancy, lactation
* patients undergoing conservative treatment for stress urinary incontinence
* ASA or other anti-platelet drug intake less than 7 days before and 7 days after procedure
* active carcinomas or status less than 5 years after treatment
* sepsis
* infection in treated region

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of patient's comfort and satisfaction | 1 year
  Improvement of patient's comfort and satisfaction measured in questionnaire ICIQ-UI SF (International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form), scale 0-21 points, higher score meaning worse outcome.
Improvement of patient's comfort and satisfaction | 1 year
  Improvement of patient's comfort and satisfaction measured in questionnaire FSFI (Female Sexual Function Index), score 2-36, higher score meaning better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Basta, PhD, Principal Investigator — Intima Clinic
Locations (1):
- Intima Clinc, Krakow, Malopolskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No